CLINICAL TRIAL: NCT01392768
Title: A Double-blind, Phase III, Multicenter, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Levetiracetam as Adjunctive Therapy, in Partial Seizures Control Associated With Refractory Focal Epilepsy
Brief Title: Efficacy and Safety of Levetiracetam in Partial Seizures Control, With or Without Secondary Generalization
Acronym: Mozart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-LPT-03(09/10)
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Epilepsy; Partial Seizures
Keywords: Epilepsy; Partial; Seizures; Adjunctive
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Oral solution (Each mL contains 100mg of levetiracetam) or immediate-release tablets (Tablets containing 500mg or 1000mg of levetiracetam)
  Arms: Levetiracetam
Drug: Placebo — Placebo, properly standardized to suit the characteristics of each dosage form (oral solution and tablets) of levetiracetam
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether levetiracetam as adjunctive therapy is effective in the treatment of partial seizures, with or without secondary generalization, associated with refractory focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 04 and 65 years, remaining the feasibility of a legal guardian in accordance with need, able to understand and provide written informed consent and able to allow compliance at the treatment and the requirements of the protocol;
* Patient´s weight ≥ 20kg;
* Consistent diagnosis of refractory focal epilepsy, with or without secondary generalization;
* Patient with onset of seizures for at least 02 years preceding the screening visit;
* Presence at least 12 partial seizures during the 03 months preceding the screening visit (04 seizures per month);

  * Only seizures that generate motor manifestation will be recorded in this study.
* Absence of brain injury progressive or expansive, previously documented by CT scan, MRI or other imaging test applicable (in the last 05 years;
* Patient with electroencephalogram performed up to 02 years before this visit;
* Subject with stable regimen (minimum of 01 month) from one to three antiepileptic drugs.

  * Vagus nerve stimulation for 04 weeks prior to V1, or use of benzodiazepines for more than 07 consecutive days will be considered as concomitant epileptic drugs)

Exclusion Criteria:

* Patients with:

  * Seizures of non epileptic origin;
  * Pseudoseizures;
  * Seizures occurring in clustered patterns (03 or more seizures in 30 minutes), in the 03 months preceding the screening visit (V1);
  * History of status epilepticus while taking antiepileptic drugs during the 03 months that preceding the screening visit (V1).
* Epileptic syndromes that occurs with cognitive deficits or secondary epilepsy evolving from some brain disease;
* History of schizophrenia or suicide attempt;
* Patients with psychiatric ill ongoing;
* Presence of severe mental retardation of any etiology;
* Previous exposure to levetiracetam;
* Women of childbearing age who had tested positive for pregnancy, or who do not use acceptable contraceptive method, or do not agree to practice reliable contraception during the study;
* Woman in pregnancy or lactation period;
* Diagnosis of renal or hepatic failure;
* Patients with genetic syndromes;
* Patient that is taking any prohibited medication (Item 9.3);
* Participation in last one year of clinical protocols, unless it can be direct benefit to subject;
* Relatives of sponsor´s or study site´s employee;
* Current evidence of clinically significant diseases: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrine, psychiatric, autoimmune, pulmonary, or another disease that block the subject participation;
* Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (e.g., blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the subject or interfere with the endpoints of study.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Partial onset seizure frequency per week. | From baseline to week 24
  Collection of seizure count throughout the whole study

SECONDARY OUTCOMES:
Safety descriptive about occurence of adverse events, evaluation of results of clinical/physical examination and ECG and laboratory tests results. | From baseline to week 30
  Collection of safety data throughout the whole study period
Proportions of response between the groups of treatment. (Responders defined as number of patients with at least 50% reduction in the number of weekly partial seizures) | From baseline to week 24
  Comparative between baseline and treatment periods
Percentage reduction from baseline in partial seizure frequency of days a week. | From baseline to week 24
  Comparative between baseline and treatment periods
Proportion of response between the groups of treatment. (Responders defined as number of subjects with at least 50% reduction in the number of days per week with partial seizures) | From baseline to week 24
  Comparative between baseline and treatment periods
Proportion between the groups of treatment without any kind of seizures. (seizure free) | 12 weeks after the titration period (period with stable regimen of the drug)
  During the evaluation period of treatment, without the titration period

CONTACTS AND LOCATIONS:
Overall Officials: Elza M Yacubian, Principal Investigator — Federal University of São Paulo